CLINICAL TRIAL: NCT04357548
Title: Optimization of Quality in Cardiopulmonary Resuscitation Through Monitor-defibrillator With Feedback System
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Principal Investigator, JOSE ANTONIO JIMENEZ HERNANDEZ, Principal investigator, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: OPTIMUMCPR
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary Resuscitation; Feedback; Quality Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Feedback system: Once the sample was selected, a test was performed in which the professionals performed 2 minutes of CPR on the dummy without any feedback system, after 5 minutes they performed 2 minutes of CPR with feedback system through the Zoll® monitor with CPR patch -D padz training, to later compare the pretest-posttest results.
  Interventions: Device: FEEDBACK

INTERVENTIONS:
Device: FEEDBACK — Once the sample was selected, a test was performed in which the professionals performed 2 minutes of CPR on the dummy without any feedback system, after 5 minutes they performed 2 minutes of CPR with feedback system through the Zoll® monitor with CPR patch -D padz training, to later compare the pretest-posttest results.

SUMMARY:
AIM: To verify the effect of a feedback system on optimizing quality during CPR on mannequins.

Hypothesis: The quality of CPR performed by healthcare professionals through a defibrillator monitor with a feedback system is higher than those that do not use a feedback system on a manikin.

METHOD Type of study: Pre-experimental with pretest-postest design. Sample: Health professionals of the General Emergency Service of the Virgen de la Arrixaca University Hospital (HCUVA).

Sampling type: Non-probabilistic for convenience. Variables: sex, age, profession, years of experience, last CPR training received, last time performing CPR, depth, frequency, quality CPR, perception of the quality of CPR.

Statistical analysis: Student's t for related samples and McNemar.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals working in the General Emergency Service of the Virgen de la Arrixaca University Clinical Hospital during the study period. They include doctors, resident doctors, and nurses.
* Health professionals from the General Emergency Service of the Virgen de la Arrixaca University Hospital who receive the training session on CPR quality and use of the defibrillator monitor with feedback system.

Exclusion Criteria:

* Health professionals who do not work in the General Emergency Service of the Virgen de la Arrixaca University Clinical Hospital during the study period.
* Health professionals who work in the General Emergency Service of the Virgen de la Arrixaca University Hospital and refuse to carry out the training and demonstration session.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects belonging to the General Emergency Department of the Hospital Clinico Universitario Virgen de la Arrixaca corresponding with doctors, resident doctors and nurses who are working in the service during the study period and receive the training session on CPR quality and the use of the defibrillator monitor with feedback system
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Depth compression | 2 minutes
  Depth of chest compressions performed by the subject
Rate compression | 2 minutes
  Frequency of the number of chest compressions per minute performed by the subject
Quality CPR | 2 minutes
  Total quality of the cardiopulmonary resuscitation performed by the subject

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Jimenez Hernandez, Doctor, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- José Antonio Jiménez Hernández, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No